CLINICAL TRIAL: NCT06877871
Title: Combined Effects of Whole Body Vibration and Abdominal Binders on Outcome Measures of Constipation in Postnatal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Iqra Ishtiaq
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Constipation in Postnatal Women; Constipation
Keywords: Constipation, C-section, pelvic floor, hemorrhoids, postpartum
MeSH Terms: conditions — Constipation; Hemorrhoids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: Whole body vibration (Experimental): WBV was developed initially for fitness and physical rehabilitation and has been moving into other areas of healthcare such as pain management and neurological recovery and improving circulation. whole body vibration (WBV) therapy for the body eases the physical functions of muscular and circulatory. Additionally, mechanical aids (e.g. abdominal binders) have been explored as support for abdominal region and proper posture, which in turn secondarily aid gastrointestinal function
  Interventions: Other: WBV utilizes mechanical vibrations to excite muscle, nerves. Abdominal binders are to help patients who have suffered abdominal trauma to stabilize core muscles, reduce pain, and improve mobility
- Experimental group: Abdominal binders (Experimental): Abdominal binders are designed primarily to help patients who have suffered abdominal trauma to stabilize core muscles, reduce pain, and improve mobility. Improved posture, better breathing and a reduction of strain on the lower back are also aided by creating gentle pressure on the abdomen. Abdominal binders are conventionally used for physical support but recent evidence supports their use in improving bowel function as increased abdominal muscle recruitment and intra-abdominal pressure, both integral to a healthy peristaltic push.
  Interventions: Other: WBV utilizes mechanical vibrations to excite muscle, nerves. Abdominal binders are to help patients who have suffered abdominal trauma to stabilize core muscles, reduce pain, and improve mobility

INTERVENTIONS:
Other: WBV utilizes mechanical vibrations to excite muscle, nerves. Abdominal binders are to help patients who have suffered abdominal trauma to stabilize core muscles, reduce pain, and improve mobility — (WBV) is a therapeutic modality that utilizes mechanical vibrations to excite muscle, nerve and tissue structures in the body. WBV was developed initially for fitness and physical rehabilitation and has been moving into other areas of healthcare such as pain management and neurological recovery and improving circulation.However, this activation can help to elevate intestinal motility, reduce bloating and help overall digestion.
  Other Names: Abdominal binders; Whole body vibrations

SUMMARY:
Constipation is a prevalent issue among postnatal women, often resulting in significant discomfort and reduced quality of life. Traditional treatments like dietary adjustments and laxatives frequently provide only temporary relief and may lead to dependency. Whole-body vibration therapy and abdominal binders have emerged as promising non-invasive interventions for improving bowel function and relieving constipation.

DETAILED DESCRIPTION:
Constipation is a complex condition arising due to many interrelated causes. Dietary inadequacies, most notably for fiber or fluid, often constitute a centerpiece of constipation. But other lifestyle factors including lack of movement and irregular bowel movements are also to blame. Known conditions affecting the gut motility, from medical perspective, include irritable bowel syndrome (IBS), diabetes, hypothyroidism, and neurological disorders including Parkinson's disease. Often listed as a side effect in medications such as opiates, antacids and antidepressants for example. Additionally, gut brain axis demonstrates that psychological aspects play a substantial part in the well being of the gut, since stress and anxiety frequently make matters worse. It is important to understand the causes of constipation to develop treatments.It is usually described as occurring less than three times per week, difficult to pass stools or passage of stools that does not feel satisfactory. Whereas, acute constipation can be often attributed to alteration in diet and water intake or stress, the chronic constipation is a long-standing pathological entity which can negatively affect the quality of life. Whole body vibration therapy (WBV) is a therapeutic modality that utilizes mechanical vibrations to excite muscle, nerve and tissue structures in the body. WBV is typically administered on a vibrating platform where the device is either controlled to deliver vibrations at specified frequencies and amplitudes as the individual performs a standing, sitting, or lying position. The vibrations produce rapid, involuntary muscle contractions- and result in a similar exercising effect without the impact to your body. Abdominal binders are conventionally used for physical support but recent evidence supports their use in improving bowel function as increased abdominal muscle recruitment and intra-abdominal pressure, both integral to a healthy peristaltic push.

ELIGIBILITY:
Inclusion Criteria:

* Females age 22-35 years
* Females underwent C-section were included in the study
* Participants who had severe constipation
* Primary gravida
* Women who had 6 months of Postpartum period
* Single fetus pregnancy

Exclusion Criteria:

* Females who had normal delivery were excluded
* History of episiotomy
* Participants taking laxative were excluded
* History of post cesarean abdominal suture infections

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Patient assessment of constipation symptoms (PAC-SYM) Questionnaire It | A total of 18 sessions were conducted over a period of 6 weeks,
  It is frequently used in clinical trials of constipation. It is an important tool for assessing the severity of patient reported symptoms of constipation. The 12-item questionnaire is divided into three symptom sub scales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe').
Patient assessment of constipation quality of life (PAC-QOL) Questionnaire | A total of 18 sessions were conducted over a period of 6 weeks,
  The PAC-QOL questionnaire is sub categorized to 4 items on physical discomfort, 8 items on psycho social discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. Response choice is a Likert scale from 0 to 4.
Modified constipation assessment scale (MCAS) | A total of 18 sessions were conducted over a period of 6 weeks,
  It is used to assess bowel function. It consists of a 3-point summated rating scale (0 = no problem ; 1 = some problem ; 2 = severe problem ) resulting in a total score that ranges from 0 ( no constipation ) to 16 ( severe constipation ).

CONTACTS AND LOCATIONS:
Overall Officials: Adeela Arif, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No